CLINICAL TRIAL: NCT05978843
Title: Comparison of Produce Prescription Benefit Dosage on Redemption
Brief Title: Comparison of Produce Prescription Benefit Dosage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A999999
Record Dates: First submitted 2023-07-17; First posted 2023-08-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Food Insecurity
MeSH Terms: interventions — Vegetables

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of three arms. Each arm will receive a different benefit amount during the 6-month intervention period, with benefit amounts determined by a percentage of the Thrifty Food Plan (TFP) - the USDA food plan used to calculate SNAP benefit rates. For ethical reasons, participants will each receive the same total benefit amount over the course of the study, with those randomized to the lower benefit arms receiving the difference between the value of the benefits issued to them and the value of the benefits issued to the highest dose group as a lump sum payment at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - 10% TFP (Active Comparator): Participants will receive $40/month in fruit and vegetable benefits for 6 months ($240 total).
  Interventions: Behavioral: Monetary benefit to purchase fruits and vegetables
- Arm 2 - 20% TFP (Active Comparator): Participants will receive $80/month in fruit and vegetable benefits for 6 months ($480 total).
  Interventions: Behavioral: Monetary benefit to purchase fruits and vegetables
- Arm 3 - 30% TFP (Active Comparator): Participants will receive $110/month in fruit and vegetable benefits for 6 months ($660).
  Interventions: Behavioral: Monetary benefit to purchase fruits and vegetables

INTERVENTIONS:
Behavioral: Monetary benefit to purchase fruits and vegetables — Participants will receive varying benefit amounts to purchase fruits and vegetables.

SUMMARY:
The goal of this study is to determine the relationship between produce prescription program 'dose' on benefit redemption, food insecurity, and fruit and vegetable consumption. Participants will be randomized to receive one of three fruit and vegetable benefit dose amounts for 6 months ($40, $80, or $110/month).

DETAILED DESCRIPTION:
Emerging evidence from the growing body of research around 'Food is Medicine' interventions shows promise that produce prescriptions (PPR) improve health by enabling purchases of healthy foods, reducing food insecurity, and improving diet quality. However, PPR amounts are often set seemingly arbitrarily, without clear connection to their intended purpose. In this study, investigators will conduct a three-armed randomized trial of 240 participants in Stockton, CA to test the impact of three 'doses' of a fruit and vegetable benefit on benefit redemption, food security, and fruit and vegetable intake. The goal of this study is to determine the relationship between PPR program 'dose' and the key intermediate outcomes of benefit redemption (primary outcome), food insecurity, and consumption of incentivized foods (secondary outcomes). Investigators will also seek to identify any 'ceiling effect' above which further increases in benefit value do not lead to further benefit redemption. This will be highly informative for subsequent PPR research. Investigators will leverage the existing infrastructure of the Vouchers 4 Veggies - EatSF produce prescription program to ensure feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Individual enrolled in a First Five Program at El Concilio California, located in Stockton, CA
* Age 18+
* English or Spanish speaking
* Literacy sufficient to complete a written survey
* Technologic capacity to complete an online survey

Exclusion Criteria:

* non English or Spanish speaking
* cognitive impairment severe enough to interfere with understanding of the survey or consent form, whether due to cognitive delay, substance abuse, dementia, mental illness, or other etiologies
* Not enrolled in a First Five Program at El Concilio California
* Actively receiving another V4V/EatSF card

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Benefit redemption | Monthly for 6 months
  Dollar amount of benefits redeemed (numerator) over total dollar amount of benefits distributed (denominator)

SECONDARY OUTCOMES:
Fruit and vegetable consumption | 0, 3, and 6 months
  Measured by NCI Dietary Screener Questionnaire (DSQ) and reported in cup-equivalents, a higher score indicates greater fruit and vegetable intake (better outcome)
Food security status | 0, 3, and 6 months
  Measured by USDA 18-item food security module. A higher score indicates more severe food insecurity (worse outcome); Scores converted to Rasch measurement scale, with a higher score indicates more severe food insecurity

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Seligman, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berkowitz SA, Baggett TP, Wexler DJ, Huskey KW, Wee CC. Food insecurity and metabolic control among U.S. adults with diabetes. Diabetes Care. 2013 Oct;36(10):3093-9. doi: 10.2337/dc13-0570. Epub 2013 Jun 11. PMID 23757436
- [Background] Bhat S, Coyle DH, Trieu K, Neal B, Mozaffarian D, Marklund M, Wu JHY. Healthy Food Prescription Programs and their Impact on Dietary Behavior and Cardiometabolic Risk Factors: A Systematic Review and Meta-Analysis. Adv Nutr. 2021 Oct 1;12(5):1944-1956. doi: 10.1093/advances/nmab039. PMID 33999108
- [Background] Seligman HK, Laraia BA, Kushel MB. Food insecurity is associated with chronic disease among low-income NHANES participants. J Nutr. 2010 Feb;140(2):304-10. doi: 10.3945/jn.109.112573. Epub 2009 Dec 23. PMID 20032485
- [Background] Ridberg RA, Bell JF, Merritt KE, Harris DM, Young HM, Tancredi DJ. Effect of a Fruit and Vegetable Prescription Program on Children's Fruit and Vegetable Consumption. Prev Chronic Dis. 2019 Jun 13;16:E73. doi: 10.5888/pcd16.180555. PMID 31198165
- [Background] Ridberg RA, Levi R, Marpadga S, Akers M, Tancredi DJ, Seligman HK. Additional Fruit and Vegetable Vouchers for Pregnant WIC Clients: An Equity-Focused Strategy to Improve Food Security and Diet Quality. Nutrients. 2022 Jun 1;14(11):2328. doi: 10.3390/nu14112328. PMID 35684128
- [Background] Stotz SA, Budd Nugent N, Ridberg R, Byker Shanks C, Her K, Yaroch AL, Seligman H. Produce prescription projects: Challenges, solutions, and emerging best practices - Perspectives from health care providers. Prev Med Rep. 2022 Aug 13;29:101951. doi: 10.1016/j.pmedr.2022.101951. eCollection 2022 Oct. PMID 36161127
- [Background] Xie J, Price A, Curran N, Ostbye T. The impact of a produce prescription programme on healthy food purchasing and diabetes-related health outcomes. Public Health Nutr. 2021 Aug;24(12):3945-3955. doi: 10.1017/S1368980021001828. Epub 2021 Apr 27. PMID 33902771